CLINICAL TRIAL: NCT03584412
Title: Feasibility Randomized-Controlled Trial of Online Acceptance and Commitment Therapy for Painful Peripheral Neuropathy in People Living With HIV: The OPEN Feasibility Study
Brief Title: OPEN Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 236730; PDF-2015-08-059 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2018-06-18; First posted 2018-07-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: HIV Neuropathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the ACT OPEN treatment condition immediately or following a 5 month wait using a 2:1 randomisation ratio (2: immediately; 1: waiting list control).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT OPEN (Experimental): Acceptance and Commitment Therapy Online for Painful Peripheral Neuropathy (ACT OPEN).
  Interventions: Behavioral: ACT OPEN
- Waiting List Control (Other): Participants in this condition will not receive any change to their usual treatment for a period of 5 months, after which they will be given access to complete the ACT OPEN treatment.
  Interventions: Other: Waiting list control

INTERVENTIONS:
Behavioral: ACT OPEN — Participants will access the ACT OPEN treatment through a secure online platform. Each session consists of brief videos and audio recordings that provide information about pain and guide participants through experiential exercises (e.g., mindfulness, values clarification, goal-setting). Participants will respond to questions assessing their experiences during the session and their progress using online messaging and/or brief telephone calls according to their preference. Therapists will provide individualised feedback. ACT OPEN consists of 12 sessions over 6 weeks. Participants will be given two further weeks to finish any uncompleted sessions, or to complete additional sessions (up to four) as agreed with their therapist.
  Arms: ACT OPEN
Other: Waiting list control — Participants will receive their usual treatment for 5 months, after which they will complete ACT OPEN as described. A waiting list control was chosen as there is no clearly credible active psychotherapy to serve as the comparator in this context, particularly in light of high drop-out rates in two previous studies of CBT for pain in HIV. Providing the online treatment without therapist support may appear to be a logical comparison group instead of a waitlist control. However, there is evidence that therapist support is a key component of online CBT and, therefore, without this support it may not represent a credible treatment against which to judge the full treatment. In the context of the feasibility aims of this trial these reasons, the use of a waiting list control is thus justified.
  Arms: Waiting List Control

SUMMARY:
The current trial will explore the feasibility of a larger efficacy trial to test a newly developed form of online CBT called Acceptance and Commitment Therapy (which we have called "ACT OPEN") for people with HIV and painful peripheral neuropathy. Participants will be recruited from HIV clinics in London, UK. Participants will be randomly chosen to receive the new ACT OPEN treatment right away or after waiting for 5 months. The treatment lasts for 8 weeks. Participants will complete self-report questionnaires to assess pain, functioning, and mood at the beginning of the study and 8 weeks and five months later.

DETAILED DESCRIPTION:
The human immunodeficiency virus (HIV) is a major health problem in the United Kingdom and worldwide. Neuropathic pain in the feet related to peripheral neuropathy is one of the most common symptoms associated with HIV. This pain is difficult to treat and medications are not effective. Chronic pain in people with HIV is related to higher levels of disability and poor quality of life.

Psychological treatments like cognitive behaviour therapy (CBT) can improve quality of life for people with chronic pain in general (not HIV-related), and there have been efforts to provide more accessible versions of CBT over the Internet. However, it is not known whether Internet-based CBT is helpful for people with HIV and chronic pain.

The current trial will explore the feasibility of a newly developed form of online CBT called Acceptance and Commitment Therapy (which we have called "ACT OPEN") for people with HIV and painful peripheral neuropathy. Participants will be recruited from HIV clinics in London, UK. Participants will be randomly chosen to receive the new ACT OPEN treatment right away or after waiting for 5 months. The treatment lasts for 8 weeks. Participants will complete self-report questionnaires to assess pain, functioning, and mood at the beginning of the study and 8 weeks and five months later.

The purpose of this study is to examine the feasibility of a larger trial evaluating the impact of online ACT for people with HIV and chronic pain in their feet. Key feasibility parameters that will be evaluated will include an estimate of the recruitment and retention rates, treatment completion rate and satisfaction, and an estimate of the effect size of changes in standard pain outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older living with HIV.
* Positive screen for peripheral sensory neuropathy, as indicated by the presence of self-reported bilateral foot pain in a symmetrical distribution (Woldeamanuel et al., 2016).
* Positive screen for symptoms of neuropathic pain in the feet, as indicated by a score of 3 or more on the patient reported outcomes section of the DN4 Neuropathic Pain Interview (Bouhassira et al., 2005; Bouhassira, Lantéri-Minet, Attal, Laurent, & Touboul, 2008)
* Pain in the feet present most days for at least 3 months.
* Average pain intensity over the past week of at least 4 on a scale from 0 (no pain) to 10 (pain as bad as you can imagine) (Zelman, Dukes, Brandenburg, Bostrom, & Gore, 2005).
* Average interference of pain with daily activities over the past 3 months is at least 4 on a scale ranging from 0 (no interference) to 10 (unable to carry on any activities) (Von Korff, Ormel, Keefe, & Dworkin, 1992).
* At least moderate symptoms of depression in the past 2 weeks, as indicated by a score of at least 10 on the PHQ-9 (Kroenke et al., 2001).

Exclusion Criteria:

* Severe symptoms of depression, as indicated by a PHQ-9 score of 23 or greater.
* Active suicidal ideation, as reflected by a score of 2 or greater on the PHQ-9 item 9 and current intent or plan to self-harm.
* A positive screen of self-reported alcohol or other substance abuse in the past 3 months as reflected by an ASSIST-Lite score of at least 3 for alcohol or at least 2 for other substances, including misuse of prescribed opioids.
* Presence of any other severe psychiatric disorder (e.g., schizophrenia, bipolar disorder, post-traumatic stress disorder) that is currently unstable or poorly controlled and likely to interfere with treatment engagement, as judged by a clinical psychologist conducting the screening.
* Currently receiving another form of regular psychotherapy (i.e., weekly appointments); involvement in psychotherapy or counselling appointments occurring less than weekly will be permitted.
* Changes to medications for mood and pain for the last 6 weeks.
* Major surgical procedure for any reason planned within the next 5 months.
* Unable to complete study procedures in English
* Unwilling to commit approximately 1-2 hours per week to complete the treatment and to do so over the Internet (note: access to a tablet/wifi will be provided for otherwise eligible participants who do not have such access; therefore, lack of internet access will not be an exclusion criterion)
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline
  Proportion of participants randomised relative to total trial referrals
Retention Rate | 8 weeks post-randomisation
  Proportion of participants who complete follow-up questionnaires
Treatment Completion Rate | 8 weeks following receipt of treatment
  We expect 70% of participants to complete at least 8/12 ACT OPEN sessions
Treatment Satisfaction | 8 weeks following receipt of treatment
  Total score on the Client Satisfaction Questionnaire (range: 8-32; higher scores reflect greater satisfaction)
Data Completeness | Baseline
  Proportion of missing items on individual questionnaires
Other Treatments Accessed | 8 weeks post-randomisation
  Self-reported frequency of use of other treatments (e.g., medical, complimentary, etc)
Patient's impression of overall change during treatment | 8 weeks following receipt of treatment
  Score on single item Patient Global Impression of Change Rating (range: 1 (very much improved) to 7 (very much worse))

SECONDARY OUTCOMES:
Pain Interference | 8 weeks post-randomisation
  Brief Pain Inventory average of pain interference subscale items score (range 0-10; higher scores reflect greater pain interference)
Social and Occupational Functioning | 8 weeks post-randomisation
  Work and Social Adjustment Scale Total Score (range: 0-40; higher scores reflect greater impairment in social and occupational functioning)
Depression Symptoms | 8 weeks post-randomisation
  PHQ-9 Total Score (range: 0-27; higher scores reflect more severe depression symptoms)
Pain Acceptance | 8 weeks post-randomisation
  Chronic Pain Acceptance Questionnaire--8 Item Version Total Score (range: 0-48; higher scores reflect greater acceptance)
Pain Intensity | 8 weeks post-randomisation
  Average of the Brief Pain Inventory pain intensity items (range: 0-10; higher scores reflect more intense pain)

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Scott, PhD, Principal Investigator — Whitney Scott
Locations (3):
- United Kingdom (3):
  - Chelsea and Westminster Hospital, London
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scott W, Guildford BJ, Badenoch J, Driscoll E, Chilcot J, Norton S, Kemp HI, Lee MJ, Lwanga J, Boffito M, Moyle G, Post FA, Campbell L, Josh J, Clift P, C de C Williams A, Rice AS, McCracken LM. Feasibility randomized-controlled trial of online acceptance and commitment therapy for painful peripheral neuropathy in people living with HIV: The OPEN study. Eur J Pain. 2021 Aug;25(7):1493-1507. doi: 10.1002/ejp.1762. Epub 2021 Mar 26. PMID 33711209